CLINICAL TRIAL: NCT02896517
Title: Support for the Rhabdomyolysis in an Emergency Department
Acronym: RHABDURGENCE
Status: Withdrawn | Type: Observational
Why Stopped: The investigator abandoned the project.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: RHABDURGENCE
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Rhabdomyolysis
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Rhabdomyolysis is a common condition in the UAA. Support is heterogeneous, it is in most cases a mass hyperhydration. The idea is to initially with an EPP simultaneously screened for the most affected by this disease and aggravating factors population, associated comorbidities.

The rhabdomyolysis prognosis depends mainly on the etiology and associated comorbidities.

* Acute renal failure and hyperkalemia are the major complications that worsen the prognosis.
* In most cases, acute renal failure is reversible. Acute renal failure caused by renal vasoconstriction with ischemia, precipitation of myoglobin in the tubules and direct cytotoxic action of myoglobin.

If the prime mover of rhabdomyolysis is ischemia (or hypoxia) cell, we now know that the tissue damage is greatly aggravated during muscle reperfusion, creating ischemia-reperfusion. Reperfusion will not only cause the release into the bloodstream of the cell contents myocytes but also an increase in necrotic areas. Indeed, the massive arrival of oxygen at the myocyte will cause significant production of free radicals, increasing their toxic effects.

Predictive factors of acute renal failure is creatinine and urea. The urine alkalinisation by bicarbonates is questionable oral alkalizing seems to be an alternative when possible (oral alkaline solution) but not used to this day.

The track N-acetyl cysteine as an antioxidant that can possibly have an effect on release of the free radicals during reperfusion by decreasing their toxicity is still not considered clinically.

DETAILED DESCRIPTION:
Main objective / secondary:

Evaluation of current professional practice:

I. Identify the most common etiologies encountered in our SAU. II. Identify the / types of people most affected by this disease III. Detect the most common complications of H0 support and evolution H48 if the patient not transferred IV. Evaluate the emergency treatment at the initial charge.

Methodology :

DESIGN:

It is a non-interventional retrospective single-center study, within the Department of Emergency GHPSJ, to an EPP and output the results regarding the type of population most affected by this disease with the most common etiologies in our support (what we are doing).

Time study:

Study on patient records being passed on to the emergency 12 months out with a diagnosis of rhabdomyolysis.

ELIGIBILITY:
Inclusion Criteria:

* All adults with CPK greater than 5N or 500 IU / L in sera to emergencies

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rhabdomyolysis admitted to the emergency department of the Hôpitel paris saint joseph
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-10-01 (Estimated); Primary Completion 2016-10-01 (Estimated); Study Completion 2016-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of patient complication by answering a questionary | Hour 0, Hour 48
  Detect the most common complications of Hour 0 support and evolution Hour 48 if the patient not transferred. Hour 0 support and evolution at Hour 48

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France